CLINICAL TRIAL: NCT03609385
Title: PRediction of Acute Coronary Syndrome in Acute Ischemic StrokE
Acronym: PRAISE
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Matthias Endres, Prof Dr med. Matthias Endres, Charite University, Berlin, Germany
Other Study IDs: EA1/057/18
Record Dates: First submitted 2018-07-06; First posted 2018-08-01 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic; Acute Coronary Syndrome
Keywords: stroke; troponin; acute coronary syndrome; culprit lesion
MeSH Terms: conditions — Ischemic Stroke; Acute Coronary Syndrome; Stroke | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients with elevated troponin: Patients with acute ischemic stroke (confirmed by cerebral imaging) and cardiac troponin values > 52 ng/l or troponin values > 14 ng/l and dynamic change > 20% will undergo coronary angiography
  Interventions: Diagnostic Test: Coronary angiography

INTERVENTIONS:
Diagnostic Test: Coronary angiography — In patients eligible for participation in the study coronary angiography, echocardiography and EKG will be performed systematically.

SUMMARY:
The primary goal of the PRAISE study is to develop a diagnostic algorithm that allows the prediction of acute coronary syndrome in stroke patients with elevated levels of cardiac troponin.

DETAILED DESCRIPTION:
Elevation of cardiac troponin can be found in about 30% of patients with acute ischemic stroke (depending on the assay used). Elevated troponin indicates increased mortality in stroke patients. There is currently little evidence regarding the ideal care of these patients. The investigators know from previous studies that approximately 25% of acute stroke patients with elevated levels of cardiac troponin have culprit lesions on coronary angiogram.

The primary goal of the PRAISE study is to develop a diagnostic algorithm that allows the prediction of acute coronary syndrome in stroke patients. To achieve this, clinical symptoms, troponin levels as well as findings on EKG, echocardiography and coronary angiography will be systematically evaluated. The PRAISE study is a multicenter study with more than 20 sites in Germany. Joint funding will be provided by DZHK (German center of cardiovascular research) und DZNE (German center of neurodegenerative diseases). Acute ischaemic stroke patients with elevated troponin are eligible for participation in the study. The primary endpoint is the diagnosis of acute coronary syndrome as established by an independent endpoint committee.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ischemic stroke based on clinical and imaging information (CT or MRI)
* diagnosis of transient ischemic attack if the initial focal neurological deficit has been examined by a neurologist and if the ABCD2-score is ≥ 4
* Elevation of high-sensitive cardiac troponins according to the rule-in/rule-out algorithm of the 2015 ESC guidelines for NSTE-ACS, i.e. highly abnormal troponin at 0 hours (> 52ng/l if hs-cTnT, Elecsys-Assay, or > 52ng/l, if hs-cTnI; Architect-Assay, or > 107 ng/l, if hs-cTnI. Dimension Vista Assay) or dynamic change > 20% of the initial value at re-test after 3 hours with at least one value above the 99th percentile of a healthy reference population
* ability to give informed consent
* onset of symptoms < 72 hours prior to hospital admission

Exclusion Criteria:

* renal insufficiency (GFR < 30 ml/min/m²)
* contraindications for coronary angiography (e.g. manifest hyperthyroidism, allergy to contrast agent)
* lesion size > 100 ml (either on Diffusion Weighted Imaging on cMRI or on CT if CT is performed > 24 hours after onset) or ASPECTS score < 7 (on CT if CT is performed < 24 hours after onset)
* Premorbid degree of dependence (mRS > 3)
* pregnancy or breast-feeding
* limited life expectancy < 1 year
* consent to participate in the study given > 72 hours after hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with acute ischemic stroke admitted to the participating sites will be systematically screened for eligibility
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Endres, Prof, Principal Investigator — Charite University, Berlin, Germany; Ulf Landmesser, Prof, Principal Investigator — Charite University, Berlin, Germany; Christian Nolte, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (28):
- Germany (28):
  - Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Charité-Campus Mitte, Berlin
  - Charité-Campus Benjamin Franklin, Berlin
  - Charité-Campus Virchow Klinikum, Berlin
  - Jüdisches Krankenhaus, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Allgemeines Krankenhaus Celle, Celle
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinikum Friedrichshafen, Friedrichshafen
  - Klinikum Fulda, Fulda
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Greifswald, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum der Ludwig-Maximilians-Universität München, Munich
  - Technische Universität München (TUM), München
  - Klinikum Nürnberg Süd, Nuremberg
  - Klinikum Osnabrück, Osnabrück
  - Universitätsmedizin Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nolte CH, von Rennenberg R, Litmeier S, Scheitz JF, Leistner DM, Blankenberg S, Dichgans M, Katus H, Petzold GC, Pieske B, Regitz-Zagrosek V, Wegscheider K, Zeiher AM, Landmesser U, Endres M. PRediction of acute coronary syndrome in acute ischemic StrokE (PRAISE) - protocol of a prospective, multicenter trial with central reading and predefined endpoints. BMC Neurol. 2020 Aug 27;20(1):318. doi: 10.1186/s12883-020-01903-0. PMID 32854663
- [Result] Nolte CH, von Rennenberg R, Litmeier S, Leistner DM, Szabo K, Baumann S, Mengel A, Michalski D, Siepmann T, Blankenberg S, Petzold GC, Dichgans M, Katus H, Pieske B, Regitz-Zagrosek V, Braemswig TB, Rangus I, Pepic A, Vettorazzi E, Zeiher AM, Scheitz JF, Wegscheider K, Landmesser U, Endres M. Type 1 Myocardial Infarction in Patients With Acute Ischemic Stroke. JAMA Neurol. 2024 Jul 1;81(7):703-711. doi: 10.1001/jamaneurol.2024.1552. PMID 38829625
- [Derived] von Rennenberg R, Litmeier S, Szabo K, Mengel A, Petersen M, Wunderlich S, Michalski D, Thomalla G, Kallmunzer B, Petzold G, Dichgans M, Siepmann T, Royl G, Ringleb PA, Nolte CH, Endres M. Cognitive performance in patients with ischemic stroke and additional myocardial injury - results from the multicenter prospective observational PRAISE study. Neurol Res Pract. 2025 Nov 4;7(1):84. doi: 10.1186/s42466-025-00446-4. PMID 41189028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stroke Patients With Elevated Troponin
Started | 254
Completed | 247
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Stroke Patients With Elevated Troponin
Number analyzed (Participants) | 247
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 75 [66 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 240
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Germany | 247

OUTCOME MEASURES:

1. Primary Outcome: Presence of Myocardial Infarction
Description: the diagnosis will be established by an independent endpoint committee
Time Frame: within seven days of admission to hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Stroke Patients With Elevated Troponin
Number analyzed (Participants) | 247
Participants
  myocardial infarction | 126
  no myocardial infarction | 121

2. Secondary Outcome: Mortality
Description: mortality will be recorded during the stay in hospital as well as after three and twelve months
Time Frame: at one week and at three and twelve months after the initial event, at 12 months reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Stroke Patients With Elevated Troponin
Number analyzed (Participants) | 247
Participants
  number of patients dead after one year | 39
  number of patients alive after one year | 208

3. Secondary Outcome: Functional Outcome
Description: functional outcome will be evaluated using the modified Rankin scale (0-6 with greater scores indicating poorer functional outcome)
Time Frame: at baseline, at one week and at three and twelve months after the initial event, 12 months reported
Population: patients with available mRS after one year
Measure: Number; unit: participants
Arm/Group | Stroke Patients With Elevated Troponin
Number analyzed (Participants) | 213
participants
  mRS 0 | 66
  mRS 1 | 35
  mRS 2 | 23
  mRS 3 | 25
  mRS 4 | 21
  mRS 5 | 4
  mRS 6 | 39

4. Secondary Outcome: Cardiovascular Events
Description: cardiovascular events include new stroke, transient ischemic attack and myocardial infarction and mortality
Time Frame: at one week and at three and twelve months after the initial event, 12 months reported
Population: participants with available follow-up data on cardiovascular events
Measure: Count of Participants; unit: Participants
Arm/Group | Stroke Patients With Elevated Troponin
Number analyzed (Participants) | 229
Participants | 60

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only severe adverse events of special interest (SAESI), i.e., MI, repeated coronary intervention, ischemic stroke or TIA, peripheral embolic artery occlusion, intracranial hemorrhage, major bleeding (type 3-5 according to BARC classification), and death were monitored for/assessed for. Other types of SAEs and Other (Not Including Serious) Adverse Events were not monitored/assessed, however, since the PRAISE study is observational and does not fall under the German Medicinal Products Act (AMG).
Arm/Group | Stroke Patients With Elevated Troponin
All-Cause Mortality (participants affected / at risk) | 39/247
Serious Adverse Events (participants affected / at risk) | 7/247
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stroke Patients With Elevated Troponin (N=247)
recurrent myocardial infarction (Cardiac disorders) | 1 (1)
ischemic stroke or TIA due to coronary angiography (Nervous system disorders) | 2 (2)
peripheral artery occlusion due to coronary angiography (Vascular disorders) | 1 (1)
major bleeding after coronary angiography (Vascular disorders) | 2 (2)
death due to coronary angiography (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03609385/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03609385/SAP_001.pdf